CLINICAL TRIAL: NCT00379951
Title: A Prospective, Multicenter, Noncomparative, Open Label Study to Evaluate the Safety, Tolerability and Efficacy of Ertapenem Sodium in the Treatment of Complicated Urinary Tract Infections
Brief Title: A Study to Assess the Safety, Tolerability and Efficacy of Ertapenem Sodium in the Treatment of Complicated Urinary Tract Infections (0826-048)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0826-048; 2006_036
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Ertapenem

ARMS (1):
- 1 (Experimental): Arm 1: ertapenem sodium
  Interventions: Drug: ertapenem sodium

INTERVENTIONS:
Drug: ertapenem sodium — ertapenem sodium as a single dose of 1gm I.V. was infused over a 30 min interval for a minimum of 3 days to a maximum of 14 days.
  Other Names: MK0826; Invanz

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of ertapenem sodium as initial therapy for the treatment of complicated urinary tract infections, including pyelonephritis in indian adults.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a complicated urinary tract infection
* Patient has acute pyelonephritis with fever, flank pain, pus in the urine, and positive urine culture
* Patient is indian and 18 years of age or greater.

Exclusion Criteria:

* Patient had a kidney transplant
* Patient had been given antibiotic therapy for condition
* Patient had poor liver function
* Patient has complete obstruction of urinary tract
* Patient has history of serious allergy to antibiotics and multivitamins
* Patient is pregnant
* Patient not likely to respond to 10 to 14 days of antibiotic therapy
* Patient not likely to survive 4 week study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2005-06; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 14 Days

SECONDARY OUTCOMES:
Compare signs and symptoms of urinary tract infections at 14 days after treatment compared with signs and symptoms before treatment | 14 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html